CLINICAL TRIAL: NCT06040905
Title: Causal Effect of Coenzyme Q10 Nutrition and Cognitive Dysfunction in the Metabolic Storm (Hyperglycemia and Sarcopenia) and Brain-derived Neurotrophic Factor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ping-Ting Lin, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CS1-22182
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Hyperglycemia; Pre-sarcopenia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Hyperglycemia | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 (Experimental): Coenzyme Q10 300 mg/day (150 mg/b.i.d.)
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Placebo (dextrin)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 300 mg/day (150mg/b.i.d)
  Arms: Coenzyme Q10
Other: Placebo — Starch, dextrin
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effect of coenzyme Q10 supplementation (150 mg/b.i.d, 300 mg/d, 12 weeks) on coenzyme Q10, glucose parameters, BDNF, myokines, and cognitive function in mild cognitive impairment (MCI) and Alzheimer's disease (AD) patients who combined with hyperglycemia but without sarcopenia, or with hyperglycemia and pre-sarcopenia.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is an aging-related disease and is considered to be a type 3 diabetes. Brain-derived neurotrophic factor (BDNF) is a potential therapeutic biomarker for AD. Studies have found that antioxidant supplementation could elevate the level of BDNF. Coenzyme Q10 is an antioxidant nutrient that participates in energy synthesis in mitochondria. Studies have shown that coenzyme Q10 has the potential to regulate blood glucose. However, there are few clinical studies to examine the effects of coenzyme Q10 supplementation on glucose and muscular metabolism and BDNF status in AD. This study will conduct an intervention study to understand the effect of coenzyme Q10 on BDNF and metabolic conditions (hyperglycemia and pre-sarcopenia) in patients with mild cognitive impairment (MCI) and AD. The study will be designed as a randomized, double-blind, cross-over, placebo-controlled study. To investigate the effect of coenzyme Q10 supplementation (150 mg/b.i.d, 300 mg/d, 12 weeks) on coenzyme Q10, glucose parameters, BDNF, myokines, and cognitive function in MCI and AD patients who combined with hyperglycemia but without sarcopenia, or with hyperglycemia and pre-sarcopenia. During the study, demographic data, mini-mental state examination, anthropometric measurements, dietary records, nutritional and muscle function assessment, quality of life, and depression assessment will be collected. Blood specimens will be also collected before and after the intervention; then the levels of coenzyme Q10, BDNF, oxidative stress, antioxidant capacity, myokines, and mitochondrial function will be analyzed. The study hopes to clarify the cause effects of coenzyme Q10 supplementation on the regulation of glucose and muscle metabolism, and cognitive function in this prospective clinical study. The results of this study will provide a reference for aging nutrition and health care.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment (MCI).
* Clinical diagnosis of Alzheimer's Disease.
* MCI and AD patients with hyperglycemia ( Fasting glucose >=100 mg/dL).
* MCI and AD patients with pre-sarcopenia (low calf circumference, low hand grip, or low muscle endurance).
* Must be able to swallow tablets.

Exclusion Criteria:

* Cancer patients.
* Severe heart, lung, liver, and kidney diseases.
* Severe disability or aphasia.
* Malnutrition (body weight changes > 5% within one month).
* Using coenzyme Q10 supplements.
* Warfarin therapy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose | 12 weeks
  Fasting glucose will measured by an automated chemistry analyzer.
HbA1C | 12 weeks
  HbA1C will measured by an automated glycated hemoglobin analyzer.
Insulin | 12 weeks
  Insulin will measured by chemiluminescence assay.
C-peptide | 12 weeks
  C-peptide will measured by chemiluminescence assay.
Brain-derived neurotrophic factor (BDNF) | 12 weeks
  Sreum BDNF level will measured by huamn BDNF ELISA kit.
Irisin | 12 weeks
  Measured by huamn Irisin ELISA kit.
Myostatin | 12 weeks
  Measured by human myostatin ELISA kit.

SECONDARY OUTCOMES:
Malondialdehyde (MDA) level | 12 weeks
  MDA will measured by thiobarbituric acid reacting substance.
Advanced Glycation End Products (AGEs) level | 12 weeks
  AGE level will measured by competitive enzyme-linked immunosorbent assay.
Total antioxidant capacity | 12 weeks
  Total antioxidant capacity will measured by a Trolox equivalent antioxidant capacity assay.
Mini-Mental State Examination (MMSE) score | 12 weeks
  The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Muscle mass | 12 weeks
  Muscle mass will measured by (Bioelectrical impedance analysis) BIA menchine.
Hand grip | 12 weeks
  Hand grip strength will be measured with a grip dynamometer.
Short Physical Performance Battery (SPPB) measurement | 12 weeks
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults. A lower score means low physical fitness.

OTHER OUTCOMES:
ATP level | 12 weeks
  ATP level will measured by ATP determination kit.
Citrate synthase level | 12 weeks
  Citrate synthase level will measured by Citrate Synthase Assay Kit.
Quality of Life in Alzheimer's Disease Measure (QOL-AD) | 12 weeks
  The QOL-AD score is the sum of all 13 items. Higher scores mean participants are more satisfied with their quality of life.
Geriatric Depression Scale (GDS) | 12 weeks
  The GDS score is the sum of all 15 items. Higher scores indicate a tendency for participants to feel depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ting Lin, Ph.D., Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No